CLINICAL TRIAL: NCT03493672
Title: Counting Steps! Integration of Objectively Assessed Physical Activity and Fitness With Smartphones in Clinical Oncology Practice.
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Laurien Maria Buffart, MD, Amsterdam UMC, location VUmc
Other Study IDs: 2017.479
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Neoplasms
Keywords: Phase I clinical trial; Phase II clinical trial; Early trial discontinuation; Objective smartphone measurements; Physical activity; Physical fitness
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Objective measurement of physical activity and fitness — Physical activity and fitness will be assessed objectively with a smartphone

SUMMARY:
Rationale:

Optimal selection of patients with cancer eligible for a clinical trial, is of utmost importance, but can be very difficult. Patients must be sufficiently fit and have a reasonable life expectancy, to be eligible for participation in clinical trials. In current clinical practice, the ECOG/WHO performance status, is used to select patients for clinical trials, and it has proven to be an independent predictor of survival in patients with cancer. This score is based on a subjective assessment of the treating physician, which can, together with the strong motivation of some patients to participate, lead to overestimation of a patient's actual physical condition and may thereby contribute to early trial discontinuation. Participation of these patients may not only harm them, but will also hamper trial conduct and outcomes.

Both, physical activity and fitness are positively associated with survival in patients with cancer. This gives rise to the investigators hypothesis that objective measurements can be of added value in the selection process. Additionally, preliminary results in 50 patients with cancer that participated in part 1 of the "Counting Steps!" project revealed that the smartphone can produce valid and reliable assessments of physical activity and fitness, and the user friendliness was rated "good" by patients.

The investigators hypothesize that measurements of physical activity and fitness with smartphones will provide more objective and accurate information about the actual physical condition of a patient with cancer.

With a better prediction of trial feasibility (without early trial discontinuation) and overall survival in patients participating in phase I-II clinical trials, the selection of eligible trial participants could be improved. In this way, it is possible to more adequately identify patients who are most likely to successfully participate in a clinical trial and thereby have the highest chance to benefit from trial participation. Successful trial participation will provide optimal palliative care to patients and improve their quality of life. In addition, it may prohibit participation of patients who are currently incorrectly included in clinical trials and suffer from toxic therapies without having a chance to benefit from treatment. A better selection of patients will be beneficial for the trial outcomes and subsequently for the development of new anticancer drugs or treatment regimens.

Objective:

The investigators aim to:

1. Identify whether objective smartphone measurements of physical activity and fitness is predictive for trial feasibility (without early trial discontinuation) in patients with cancer participating in phase I-II clinical trials.
2. Evaluate the feasibility and acceptability of the use of the smartphone's objective assessments of physical activity and fitness in clinical practice.

Study design: Observational study

Study population:

• 135 patients with hematologic or solid cancer referred to the VU medical center for participation in phase I-II clinical trials.

Intervention:

In this observational study, patients will not receive an additional intervention.

Main study parameters/endpoints:

Prior to the start of medical treatment, physicians will rate the performance status, and participants will wear a smartphone for one week to measure the daily number of steps, to complete the 6 minute walk test using the smartphone application, and to fill out the 5-item physical function subscale of the EORTC QLQ-C30. These assessments will be repeated after 4 and 8 weeks.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

No extra visits to the hospital will be necessary. Participation in this study will not cause any additional risks or expected benefits for participants. It will only deliver knowledge, which may be used in the future to better select patients eligible for participation in phase I-II clinical trials or even for regular treatment. Participation in the study will only cost time for patients. The patients will be asked to wear a smartphone for a week, have to perform a six-minute walk test (6MWT) once in this week and have to complete a questionnaire about their own physical function once. Subsequently, patients will repeat those measurements 4 and 8 weeks after inclusion in the phase I-II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer, referred for treatment in phase I/II clinical trial
* Written informed consent

Exclusion Criteria:

* Already started treatment in phase I/II clinical trial
* Inability to understand the Dutch language
* Cognitive disorders or severe emotional instability
* Reasons why mobilizing is impossible, like fracture, paraplegia etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with advanced cancer referred to the outpatient department of Medical Oncology and Hematology of the VU medical center, for treatment in a phase I/II clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Early trial discontinuation | 2 months
  Early trial discontinuation is defined as discontinuation of trial in the first two months after inclusion, dichotomized into yes or no

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival is defined as the time between start of trial participation and death of any cause and will be tracked via the registration of the original clinical trial
Progression free survival | 1 year
  Progression free survival is defined as the time between trial participation and the clinically or radiologically confirmation of progressive disease (established via RECIST-criteria) as defined by the original clinical trial and will be tracked via the registration of the original clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided